CLINICAL TRIAL: NCT03982901
Title: Effect of Mental Stress on Myocardial Perfusion and Myocardial Blood Flow in Women With Chest Pain and Coronary Artery Stenosis Less Than 50%
Brief Title: Effect of Mental Stress on Myocardial Perfusion in Women
Acronym: MS in women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019298H(R3)
Record Dates: First submitted 2019-06-02; First posted 2019-06-12 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2020-08

CONDITIONS: Non-Obstructive Coronary Atherosclerosis
Keywords: Stress; Ischemia; PET-CT
MeSH Terms: conditions — Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- women with chest pain (Experimental): women with chest pain and coronary artery stenosis less than 50%
  Interventions: Diagnostic Test: Mental Stress Test
- healthy women (Sham Comparator): women without chest pain and coronary artery stenosis less than 50%
  Interventions: Diagnostic Test: Mental Stress Test

INTERVENTIONS:
Diagnostic Test: Mental Stress Test — In this study, we compare MSIMI prevalence in the two groups (chest pain group and no chest pain group). Each subject in both groups receive the same mental stress test process, and the mental stress test process have 3 consecutive stress tests, which including: Stroop Color-Word test; Public speaking with anger recall test and Mental arithmetic test.

SUMMARY:
Mental stress-induced myocardial ischemia(MSIMI) has been recognized a significant clinical problem. Evidence has shown that individuals with MSIMI have 2 to 2.5 times higher risk to develop a major averse cardiovascular events over 3-5 years, compared to their counterparts who have no MSIMI. Nevertheless, investigations into the study of MSIMI among women who have chest pain but artery stenosis < 50% have been lacking. In this project, the investigators used positron emission tomography (PET) to evaluate perfusion defect during mental stress to diagnose MSIMI. Women with chest pain and coronary artery stenosis < 50% were included as the experimental group, age-matched healthy people as the control group, the aim of this study is to compare the incidence of MSIMI in the two groups. At the same time, the study also observe the change of MBF during mental stress and the relationship between MBF and MSIMI.

DETAILED DESCRIPTION:
The goals of this project are to assess MSIMI prevalence in chest pain women with coronary artery stenosis less than 50%, as compared to age matched healthy women, and the MBF change during mental stress and adenosine vasodilator stress by PET with N-13 ammonia . This study will also establish the methodology of echocardiography to diagnose MSIMI by comparing with PET. To evaluate the consistency of myocardial blood flow (MBF by PET-CT) and peripheral blood flow (PAT ratio by EndoPAT) during stress test. and to explore the pathogenesis of MSIMI from aspects of neuroendocrine mechanism, sex hormone level, humoral immunity index and proteome expression.

The stress testing will be conducted at the PET-CT and echocardiography unit of Guangdong Provincial People's Hospital. Following a 20-minute calibration-rest period, participants will be asked to complete a series of 3 consecutive mental stress tasks. The mental stress tests are embedded in the virtual reality device, and the subjects can carry out the mental stress test with the virtual reality device on their heads. (1) Stroop Color-Word test, is administered by computer on a video monitor. A word appeared in the middle of the screen-Red, Green, Yellow, or Blue-in one of these four colors. At the bottom of the screen the words Red, Green, Yellow, and Blue appeared with the font color not matching the word meaning. The participant is asked to match the color of the word in the middle of the screen with the meaning of the color word at the bottom by clicking on the correct option, which lasts about 4 minutes. and then (2) Public speaking with anger recall: during this test, patients will be asked to give a speech on a recent situation in which they experienced anger to an audience of three observers (doctors) after 1 minute of preparation. Prior to the speech, subjects are told that their speech will be evaluated on their description of the situation, as to what happened, what they thought, felt, what they did, and what happened as a result. If they run out of things to say, the research tech will prompt them with questions to elicit more content until the three minutes are up. and at last the (3) Mental arithmetic: during this test, patients will be asked to perform a series of serial subtractions beginning at a given number which will be different for each repeated test and will be chosen by the tester from a fixed list of various numbers, with encouragement to perform calculations as quickly as possible; Each mental stress lasts for 4 minutes, there is no rest between the two mental stress, and the whole process of mental stress is 12 minutes.

ELIGIBILITY:
The inclusion criteria are as follows:

1) Women with chest pain and coronary artery stenosis < 50% 2) Participate in the trial voluntarily and sign the informed consent form; 3) older than 18 and less than 75 years old, female; 4) be able to cooperate with the completion of evaluation and inspection. Exclusion criteria.

1. Chest pain caused by diseases other than the cardiovascular system such as Aortic dissection, Pulmonary embolism;
2. Combined with pulmonary embolism;
3. Combined with aortic dissection;
4. A serious life-threatening arrhythmias;
5. Combined with cardiomyopathy or severe valvular disease;
6. New York Heart Association(NYHA) class IV;
7. Recent myocardial infarction within 1 month;
8. Combined with severe mental illness, such as schizophrenia, Active suicidal ideation etc.
9. History of substance and alcohol abuse in the previous 12 months;
10. Significant cardiac, pulmonary, metabolic, renal, hepatic disease, or malignancy, interfering with patient's participation in this study;
11. Currently taking antidepressant or antianxiety medications within 1 month;
12. Participated in other clinical trials within 3 months;
13. Cognitive impairment or inability to cooperate with researchers.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2019-06-18 (Actual); Primary Completion 2021-04-29 (Actual); Study Completion 2021-04-29 (Actual)

PRIMARY OUTCOMES:
MSIMI (Measures as perfusion deficit with mental stress test via PET-CT) prevalence in chest pain women with coronary artery stenosis less than 50%, as compared to age matched healthy women. | half an hour
  Percentage of participants wih an presence of mental stress-induced myocardial ischemia (MSIMI) during the 3 mental stressors.
  MSIMI is defined by the following: compared to rest, 1) Each myocardial segment was scored from 0 to 4, with 0 being normal, 1 possibly normal, 2 definitely abnormal, 3 severely abnormal, and 4 no perfusion. The investigators calculated summed scores in a conventional fashion, including a summed stress score, a summed rest score, and a summed difference score. A summed difference score ≥3 is typically used as evidence of MSIMI.
The MBF change during mental stress test | half an hour
  The MBF change during mental stress test

SECONDARY OUTCOMES:
Blood flow reserve in women with chest pain and coronary artery stenosis < 50% . | half an hour
  Bood flow reserve of participants using Adenosine
The consistency of PET-CT myocardial scanning and color Doppler echocardiography (contrast echocardiography, spot tracking) for the diagnosis of MSIMI. | 30 days
  The consistency between PET-CT and Doppler echocardiography (contrast echocardiography, spot tracking) in diagnosing MSIMI
The consistency of myocardial blood flow (MBF by PET-CT) and peripheral blood flow (PAT ratio by EndoPAT) under pressure test. | 2 hours
  The consistency between myocardial blood flow and peripheral blood flow during mental stress test
The neuroendocrine change in MSIMI(+) group, as compared with MSIMI(-) group. | 1 hour
  The cause of MSIMI
The difference of sex hormone level between MSIMI(+) group and MSIMI(-) group | 1 hour
  The cause of MSIMI
The difference of humoral immunity index level between MSIMI(+) group and MSIMI(-) group. | 1 hour
  The cause of MSIMI
The difference of proteome expression level between MSIMI(+) group and MSIMI(-) group. | 2 days
  The cause of MSIMI

CONTACTS AND LOCATIONS:
Overall Officials: Qingshan Geng, Study Chair — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
All data (including data dictionaries) from individuals consent to the present project, after de-identification, will be shared that include all been discussed in this article. Study protocol, statistical analysis plan, and analytic code are available for sharing. We anticipate data sharing will be ready 6 months after the publication of the primary end point of this project, and ending 36 months following article publication. Our data may be shared with investigators who provide a methodologically sound proposal with approval of an independent review committee. Proposals should be directed to gengqsh@163.net. To gain access, data requestors will need to sign a data access agreement with our institution. Data are available for 5 years at the data management center.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Derived] Liu Y, Jiang W, Wang H, Xu M, Liao Y, Zhou H, Bai B, Liu F, Yin H, Liu Q, Liang Y, Yu X, Guo L, Wang S, Ma H, Geng Q. Objective Ischemia, Subjective Angina, and Psychological Distress in Angina With No Obstructive Coronary Disease. J Am Heart Assoc. 2024 Aug 6;13(15):e034644. doi: 10.1161/JAHA.124.034644. Epub 2024 Jul 31. PMID 39082421
- [Derived] Ma H, Guo L, Fei H, Yin H, Wang H, Bai B, Liu Y, Wang S, Geng Q, Jiang W. Assessing mental stress on myocardial perfusion and myocardial blood flow in women without obstructive coronary disease: protocol for a mechanistic clinical trial. BMJ Open. 2020 Dec 8;10(12):e038362. doi: 10.1136/bmjopen-2020-038362. PMID 33293388